CLINICAL TRIAL: NCT00571714
Title: Comparison of Standard Therapy,Peginterferon Alpha-2a + Ribavirin for 48 Weeks VS Peginterferon Alph-2a + Ribavirin + Betaine for 12 Weeks Followed by 36 Weeks Standard Therapy in Untreated Adults With Chronic Hepatitis C Genotype 1
Brief Title: Pilot Comparison of Standard Antiviral Therapy With and Without 12 Weeks of Betaine in Genotype 1 Naive Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0159-07-FB
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Pilot Comparison; Peginterferon alph-2a; Ribavirin; Betaine; Genotype 1; Treatment naive
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a; Betaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Standard Peginterferon alpha-2a plus Rivavirin Therapy (Active Comparator): Peginterferon alpha-2a once a week plus weight based ribavirin (800-1400mg/day)in 2 divided daily doses
  Interventions: Drug: Peginterferon alpha-2a and ribavirin
- 2 Peginterferon alpha-2a plus Rivavirin Therapy with Betaine for First 12 Weeks (Active Comparator): Peginterferon alpha-2a once a week plus weight based ribavirin (800-1400mg/day) in 2 divided daily doses plus betaine (20gm/day) in 2 divided doses for 12 weeks followed by Peginterferon alpha-2a q week plus weight based ribavirin (800-1400mg/day) in 2 divided daily doses for 36 weeks
  Interventions: Drug: Peginterferon alpha-2a , ribavirin and betaine

INTERVENTIONS:
Drug: Peginterferon alpha-2a and ribavirin — Peginterferon alpha-2a 180mcg by subcutaneous injection every week and weight based ribavirin, 800 to 1400mg/day by mouth in two divided doses every day for 48 weeks
  Other Names: Pegasys; Copegus
  Arms: 1 Standard Peginterferon alpha-2a plus Rivavirin Therapy
Drug: Peginterferon alpha-2a , ribavirin and betaine — Peginterferon alpha-2a 180mcg given by subcutaneous injection every week plus weight based ribavirin 800 to 1400 mg/day by mouth in divided doses twice a day plus betaine 10 gm dissolved in juice twice a day for twelve weeks followed by peginterferon alpha-2a 180 mcg given by subcutaneous injection every week plus weight based ribavirin 800 to 1400mg/day by mouth in divided doses twice a day for 36 weeks.
  Other Names: Pegasys; Copegas
  Arms: 2 Peginterferon alpha-2a plus Rivavirin Therapy with Betaine for First 12 Weeks

SUMMARY:
The primary purpose of the study is to compare the safety and effectiveness of standard treatment for chronic hepatitis C using peginterferon alpha-2a (Pegasys) and ribavirin (Copegus) to those same medications plus a dietary supplement called betaine when added for the first 12 weeks of treatment.

Peginterferon alpha-2a (Pegasys) and ribavirin (Copegus) are approved by the FDA (Food and Drug Administration) for the treatment of chronic hepatitis C.

Betaine is a dietary supplement and occurs naturally in the body. It is not a medication regulated by the FDA or an approved drug for chronic hepatitis C.

DETAILED DESCRIPTION:
Although pegylated alpha interferon and ribavirin will likely be part of the core therapy for chronic HCV for the next several years, there are a number of complimentary antiviral agents in development including protease or polymerase inhibitors, RNA vaccines and immunomodulators (5). However, it would be unlikely to have FDA approval for any of these newer agents before the next 3 - 5 years, i.e. 2010-2012.

Betaine, a naturally occurring anti-oxidant metabolite of choline and an amino acid analog (tri-methyl-glycine), serves as a methylation agent to re-methylate damaged cell proteins or enzymes (6). By virtue of its metabolic role in decreasing toxic metabolites, betaine also protects against alcohol-induced fatty liver and apoptosis. Recently, pilot studies performed both at the Mayo Clinic and here at UNMC showed its applicability as a treatment of non-alcoholic fatty liver in human subjects (7, 8).

Betaine has also recently been found to promote interferon function by overcoming HCV - induced inhibition of interferon signaling (9). Naturally-occurring HCV proteins during human infection can hypo-methylate proteins integral to the Jak - STAT (signal transducers and activators of transcription) pathway, thereby inhibiting the antiviral activity of interferon. In cultured cells betaine administration, in a physiologically attainable concentration, restored STAT methylation and improved interferon signaling (9).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be willing to give informed consent and be able to adhere to dose and visit schedules.
* History of chronic hepatitis C as documented by either anti-HCV or HCV RNA positivity.
* Adult subjects 19-70 years of age, of either gender
* Liver biopsy within 3 years prior to the screening 1 visit.
* Compensated liver disease with the following maximum hematologic, biochemical and serologic criteria at the Screening visit (WNL=within normal limits) Hemoglobin > 12 g/dl for females and >13 g/dl for males, WBC > 3000/mm3, Platelets > 80,000/mm3, Direct Bilirubin - WNL. Indirect bilirubin - WNL, Albumin - WNL, Serum Creatinine - WNL.
* Fasting glucose should be 70 -140 mg/dl, results between 116-140 require a HbA1c < 8.5%
* TSH - WNL
* Subjects with a history of mild depression may be considered for entry in to this study provided that a pretreatment assessment of the subject's affective status supports that the subject is clinically stable.
* Subjects with a history of substance abuse must have abstained from using the substance for at least one year prior to the Screening visit.
* Antinuclear antibodies (ANA) < 1:320
* No radiologic evidence of a focal mass suggestive of hepatoma and/or ascites.

Exclusion Criteria:

* Pregnant or nursing subjects. Subjects who intend to become pregnant during the study period. Subjects with partners who intend to become pregnant during the study period.
* History of new hepatitis C exposure within the last 6 months
* Prior treatment for chronic hepatitis C.
* Current or intended use of G-CSF and/or GM-CSF during the stud period is prohibited. Current use of erythropoietin (EPO) is prohibited.
* Suspected hypersensitivity to any interferon product or ribavirin
* Participation in any other clinical trial within 30 days of Screening visit
* Treatment with any investigational drug within 30 days of Screening visit 1.
* Any other cause for liver disease other than CHC.
* Coagulopathies including hemophilia
* Hemoglobinopathies
* G6PD deficiency
* Coinfection with HIV and/or HBV
* Evidence of active or suspected malignancy or a history of malignancy within the last five years (with the exception of adequately treated basal cell carcinoma of the skin).
* Evidence of decompensated liver disease such as history or presence of ascites, bleeding varices or hepatic encephalopathy
* Subjects with organ transplants other than cornea or hair transplant
* Any Known preexisting medical condition, that could interfere with the subject's participation in and completion of the study.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2010-03-04 (Actual); Study Completion 2010-03-04 (Actual)

PRIMARY OUTCOMES:
Sustained Viral Response 24 weeks following the end of anti-viral therapy | 72 weeks
  no patients enrolled

SECONDARY OUTCOMES:
Comparison of rapid and early virologic response in the first 4 and 12 weeks of therapy | 12 weeks
  no patients enrolled
Comparison of the safety of the two treatment regimens | 48 weeks
  no patients enrolled
Comparison of ALT normalization between the two regimens | 48 weeks
  no patients enrolled
Comparison of the effect on interferon gene signaling in peripheral blood mononuclear cells between the two regimens in the first 12 weeks of therapy. | 12 weeks
  no patients enroll

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Mailliard, MD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No
no patients enrolled to the study

REFERENCES:
- [Background] Abdelmalek MF, Angulo P, Jorgensen RA, Sylvestre PB, Lindor KD. Betaine, a promising new agent for patients with nonalcoholic steatohepatitis: results of a pilot study. Am J Gastroenterol. 2001 Sep;96(9):2711-7. doi: 10.1111/j.1572-0241.2001.04129.x. PMID 11569700
- [Background] Duong FH, Christen V, Filipowicz M, Heim MH. S-Adenosylmethionine and betaine correct hepatitis C virus induced inhibition of interferon signaling in vitro. Hepatology. 2006 Apr;43(4):796-806. doi: 10.1002/hep.21116. PMID 16557551
- [Result] 8. Mukherjee S, Bernard T, Schafer D, et al. Impact of betaine on hepatic fibrosis and homocysteine in nonalcoholic steatohepatitis: a prospective cohort study [abstract]. Hepatology 2005; 42: 610A.